CLINICAL TRIAL: NCT04297787
Title: Safety and Efficacy of Thrombolysis in Combination With Endhole Aspiration in the Treatment
Brief Title: Safety and Efficacy of Thrombolysis in Combination With Endhole Aspiration in the Treatment of Acute DVT
Acronym: INDIGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00145734
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Acute Deep Vein Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): The treatment protocol the study team will be following is as follows for all enrolled patients. First, a pulse spray tPA infusion with 20 cc of 8 mg tPA and saline will be administered to the thrombus with a 20-minute dwell time. Afterwards, an 8F curved sheath (Indigo 8 Torq Tip, ranges 85 to 115 cm) with CAT8 penumbra device will be used to aspirate the thrombus. If the operating physician deems necessary, they will have the option at that point to balloon plasty, stent, or use catheter-directed thrombolysis at this point. Clinical parameters such as areas of clinically-significant stenosis, extent of thrombus, (more parameters) will be tracked at the time of the procedure. The device is being used is FDA approved and being used according to FDA indications.
  Interventions: Device: Thrombolysis in combination with endhole aspiration

INTERVENTIONS:
Device: Thrombolysis in combination with endhole aspiration — The treatment protocol the study team will be following is as follows. First, a pulse spray tPA infusion with 20 cc of 8 mg tPA and saline will be administered to the thrombus with a 20-minute dwell time. Afterwards, an 8F curved sheath (Indigo 8 Torq Tip, ranges 85 to 115 cm) with CAT8 penumbra device will be used to aspirate the thrombus. If the operating physician deems necessary, they will have the option at that point to balloon plasty, stent, or use catheter-directed thrombolysis at this point. Clinical parameters such as areas of clinically-significant stenosis, extent of thrombus, (more parameters) will be tracked at the time of the procedure. The device is being used is FDA approved and being used according to FDA indications.

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of thrombolysis in combination with endhole aspiration in the treatment of acute deep vein thrombosis (DVT). Secondarily, the study team hope to illuminate the financial implications of single session catheter directed therapy versus a potential 48 hour lysis procedure (Lysis is an approach in which vascular specialists deliver clot-dissolving drugs directly to the site of the clot through a catheter).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Onset of acute DVT occurred <14 days
* Ability to undergo thrombolysis in combination with Indigo endhole aspiration device

Exclusion Criteria:

* Under 18 years of age
* Presence of subacute (14-28 days) or chronic DVT (>28 days)
* Contraindication to mechanical thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Post-thrombotic Syndrome (PTS) severity using the Villalta score | 1 month
  Patient outcomes will be measured through clinical grading of PTS severity using the Villalta score, a clinical measure for the post-thrombotic syndrome that grades the severity, from 0 (absent) to 3 (severe), of each of 5 patient-rated symptoms (pain, cramps, heaviness, pruritus, and paresthesia) and 6 clinician-rated clinical signs (edema, redness, skin induration, hyperpigmentation, venous ectasia, and pain of calf). A summative score of 5 or more on the Villalta scale indicates the presence of the postthrombotic syndrome (Villalta).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Rohr, MD, Principal Investigator — Interventional Radiology-Vascular
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No